CLINICAL TRIAL: NCT07216846
Title: The Geriatric Emergency Department Pharmacologic Harm Prevention Project
Acronym: GREAT PHARM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Responsible Party: Principal Investigator, Richard Shih, Principal Investigator, MD, Florida Atlantic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2505160
Record Dates: First submitted 2025-10-09; First posted 2025-10-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Fall; Fall Accident; Poly Pharmacy; Adverse Drug Events; Pharmacogenomic Drug Interaction; Pharmacogenomic Testing
Keywords: Fall; Geriatric; Pharmacogenomic; adverse drug event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacogenomic-Guided Prescribing pathway (Experimental): Pharmacogenomic test results will be transmitted to the participant's primary care physician to support medication optimization and prescribing decisions. Follow-up assessments will be conducted by telephone approximately 14 days after enrollment and then monthly for six months. These structured interviews will capture information on falls, fall-related injuries, medication changes, adverse drug effects, and new medical conditions.
  Participants will also complete a monthly calendar to document medication changes, falls, and fall-related injuries. Medical records from the participant's primary care physician will be reviewed for corroborating information on falls, fall-related injuries, medication changes, medication-related side effects, and newly diagnosed medical problems.
  Interventions: Other: DNA care pathway
- Emergency Department care pathway ---control (No Intervention): Participants randomized to the current Emergency Department care pathway will continue to receive standard prescribing practices without immediate use of pharmacogenomic results. Follow-up assessments will occur by telephone approximately 14 days after enrollment and then monthly for six months. These calls will collect data on falls, fall-related injuries, medication changes, adverse drug effects, and new medical conditions.
  Participants will also complete a monthly calendar documenting medication changes, falls, and fall-related injuries. Medical records from the participant's primary care physician will be reviewed to identify additional falls, injuries, medication changes, side effects, and new medical problems. At the conclusion of the study, pharmacogenomic testing results will be provided to the participant's primary care physician to support future prescribing decisions.

INTERVENTIONS:
Other: DNA care pathway — Pharmacogenomic test results will be transmitted to the participant's primary care physician to support medication optimization and prescribing decisions. Follow-up assessments will be conducted by telephone approximately 14 days after enrollment and then monthly for six months. These structured interviews will capture information on falls, fall-related injuries, medication changes, adverse drug effects, and new medical conditions.
  Participants will also complete a monthly calendar to document medication changes, falls, and fall-related injuries. Medical records from the participant's primary care physician will be reviewed for corroborating information on falls, fall-related injuries, medication changes, medication-related side effects, and newly diagnosed medical problems.
  Arms: Pharmacogenomic-Guided Prescribing pathway

SUMMARY:
The goal of this project is to determine whether pharmacogenomic testing (using participants' DNA) can help optimize medication prescribing and reduce side effects in older adults taking five or more medications.

The main questions it aims to answer are:

* Can DNA-based prescribing reduce medication-related side effects, especially falls and fall-related injuries?
* Does providing pharmacogenomic results to primary care physicians improve medication safety compared with usual care?

Researchers will compare two groups:

1. DNA Care Pathway: Physicians receive patients' DNA results to guide prescribing.
2. Emergency Department Care Pathway: Physicians provide usual care; DNA results are shared only after study completion.

Participants will:

* Provide a cheek swab sample for DNA analysis (1 minute).
* Receive monthly follow-up phone calls for 6 months to track falls, injuries, medication changes, and side effects.
* Complete a fall and medication calendar.
* Allow researchers to review primary care physician medical records for study outcomes.

Approximately 1,000 participants will take part, with follow-up lasting about 6-7 months.

DETAILED DESCRIPTION:
Background and Rationale Medication prescribing is one of the most common medical interventions. In the U.S., 81% of adults report taking at least one medication in the past week, and 50% take prescription medications. Among older adults, 39% meet the criteria for polypharmacy, defined as the use of five or more chronic medications.

Polypharmacy is strongly associated with adverse drug events (ADEs). Each day, approximately 750 older adults in the U.S. are hospitalized due to ADEs, with half of these patients taking five or more medications. Nearly 60% of older adults are prescribed at least one potentially unnecessary medication.

Traditional prescribing often follows a "one-size-fits-all" approach, which does not account for genetic differences in how individuals metabolize drugs. These genetic variations can lead to ineffective treatment or harmful side effects. Pharmacogenomic-guided prescribing may provide a safer, more personalized approach by identifying drug-gene interactions and tailoring medication choices.

Falls and Medication Safety Falls are one of the most serious and preventable ADEs among older adults. Falls are the leading cause of injury-related morbidity and mortality in older populations, with over 700,000 hospital falls in the U.S. annually. Polypharmacy, especially the use of fall-risk-increasing drugs (FRIDs), contributes substantially to this problem.

By integrating pharmacogenomic testing into medication management, clinicians may be able to reduce fall-related ADEs and improve overall prescribing safety.

Study Objectives and Aims The Geriatric Emergency Department Pharmacologic Harm Prevention Project (The GREAT PHARM) seeks to evaluate whether pharmacogenomic-guided prescribing can reduce ADEs and falls among older adults.

Aim 1: Compare the incidence of recurrent falls, ADE-related emergency department (ED) visits, and all-cause mortality in patients receiving pharmacogenomic-guided medication optimization versus usual care.

Secondary Aim 1: Assess barriers to implementing pharmacogenomic-based prescribing. Aim 2: Determine the prevalence of harmful gene-drug interactions and abnormal drug levels in older adults presenting to the ED after a fall.

Aim 3: Compare self-reported wellbeing and health satisfaction between patients who receive pharmacogenomic-guided prescribing and those receiving usual care.

Study Design

* This is a randomized clinical trial enrolling approximately 1,000 participants aged 65 and older.
* Eligibility: Adults ≥65 years presenting to the ED with a ground-level fall.
* Exclusion criteria: Hospice care or Do Not Resuscitate (DNR) status.

Randomization: Participants will be randomized (via REDCap) into two study arms:

1. Control Group (Current Care) - Standard prescribing practices; pharmacogenomic results provided to primary care physicians only after study completion.
2. Intervention Group (Pharmacogenomic-Guided Prescribing) - Standard care plus pharmacogenomic results provided to the primary care physician during the study for medication optimization.

Interventions

All participants will:

* Provide a one-time cheek swab sample for DNA analysis (testing 26 metabolic enzyme systems).
* If blood is drawn for routine ED care, provide an additional small blood sample (~5cc) for drug-level analysis. Blood concentrations will be assessed using mass spectrometry at the Florida Atlantic University Bioanalytical Core Facility.
* Complete a monthly calendar to record medication changes, falls, and fall-related injuries.
* Participate in monthly follow-up phone calls (for 6-7 months) to track falls, side effects, and overall health.
* Authorize access to primary care physician medical records for up to one year to confirm study outcomes.

Outcome Measures

Primary Outcomes:

1. Incidence of recurrent falls during 6-7 months of follow-up.
2. Incidence of ADE-related ED visits.
3. All-cause mortality.

Secondary Outcomes:

1. Prevalence of harmful gene-drug interactions in older adults presenting with falls.
2. Prevalence of abnormal drug levels in patients with pharmacogenomic variations.
3. Patient-reported wellbeing and health satisfaction.
4. Barriers to implementation of pharmacogenomic-guided prescribing.

Duration of Participation Each participant will be followed for approximately 6-7 months, with ongoing monitoring through phone calls, calendars, and medical record review.

Significance This trial will evaluate whether personalized prescribing guided by DNA testing can reduce medication-related harm, prevent recurrent falls, and improve overall quality of life for older adults. If successful, the study will provide strong evidence for integrating pharmacogenomic-guided prescribing into standard clinical care for geriatric patients at risk of medication-related harm.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 65 with a ground level fall

Exclusion Criteria:

* hospice and/or DNR status.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent falls -self reported and chart review | 6-7 months
  Incidence of recurrent falls during 6-7 months of follow-up. Around the fourteenth day of the study and then once a month for the following six months, participants will receive a follow-up phone call to assess any falls that may have occurred. In addition, each participant will receive a calendar to record falls during the month. At six-month, the primary care physician medical records will be reviewed to check for any additional falls.
Incidence of ADE-related ED visits- self reported and chart review | Time Frame: 6-7 months
  Incidence of ADE-related ED visits during 6-7 months of follow-up. Around the fourteenth day of the study and then once a month for the following six months, participants will receive a follow-up phone call to assess any ADE-related ED visits that may have occurred. At six-month, the primary care physician medical records will be reviewed to check for any additional ADE-related ED visits.
All-cause mortality - Florida Death Registry | Time Frame: 6-7 months
  During 6-7 months of follow-up. All participants will be cross-referenced with the Florida Death Registry to identify mortality outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Richard Shih, MD, Principal Investigator — Florida Atlantic University
Locations (1):
- Delray Medical Center, Delray Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to do it